CLINICAL TRIAL: NCT06004921
Title: A Phase 1, Double-Blinded, Randomised, Placebo-Controlled, Single Ascending Dose (SAD) Study in Healthy Subjects to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of AB801
Brief Title: A Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of AB801 in Healthy Volunteers
Acronym: ARC-26
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ARC-26
Record Dates: First submitted 2023-08-15; First posted 2023-08-22 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-05

CONDITIONS: Cancer
Keywords: AB801; Healthy volunteer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1 - AB801 Dose A (Experimental): Participants will receive a single dose of AB801 or placebo
  Interventions: Drug: AB801; Drug: Placebo
- Cohort 2 - AB801 Dose B (Experimental): Participants will receive a single dose of AB801 or placebo
  Interventions: Drug: AB801; Drug: Placebo
- Cohort 3 - AB801 Dose C (Experimental): Participants will receive a single dose of AB801 or placebo
  Interventions: Drug: AB801; Drug: Placebo
- Cohort 4 - AB801 Dose D (Experimental): Participants will receive a single dose of AB801 or placebo
  Interventions: Drug: AB801; Drug: Placebo

INTERVENTIONS:
Drug: AB801 — Administered as specified in the treatment arm
Drug: Placebo — Administered as specified in the treatment arm

SUMMARY:
The primary purpose of this study is to determine the safety and tolerability of AB801, and to understand the pharmacokinetic (PK) profile of AB801 when taken as a capsule and tablet in healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy as determined by medical evaluation by study physician
* Body mass index (BMI) of 18.0 to 32.0 kilogram (kg)/meter (m)^2 as measured at screening
* Weight ≥ 50 kg at screening
* Must agree to adhere to the protocol defined contraception requirements

Key Exclusion Criteria:

* Do not have suitable veins for multiple venepunctures/cannulation as assessed by the study physician
* Prolonged QT interval defined as mean Corrected QT interval by Fridericia's formula (QTcF) ≥ 450 msec for males and > 470 millisecond (msec) for females at screening and pre-dose
* Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the study physician
* Received any study medicine in a clinical research study within the last 90 days
* Taking, or have taken, any prescribed or over-the-counter drugs including gastric acid reducing agents and including CYP3A inhibitor and/or inducers

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-02-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 30 days
Area Under the Plasma Drug Concentration-Time Curve (AUC) | Predose, Up to 120 hours postdose
Maximum Concentration (Cmax) in Plasma | Predose, Up to 120 hours postdose
Time to Maximum Concentration (Tmax) in Plasma | Predose, Up to 120 hours postdose
Half-Life Time (t1/2) | Predose, Up to 120 hours postdose

SECONDARY OUTCOMES:
Change from Baseline in Holter Electrocardiogram Monitoring Scale | Predose up to 25 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (1):
- Quotient Sciences - Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy